CLINICAL TRIAL: NCT00004147
Title: A Phase I/II Study of Col-3 Administered on a Continuous Daily Oral Schedule in Patients With Recurrent High-Grade Astrocytoma
Brief Title: COL-3 in Treating Patients With Progressive or Recurrent Brain Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067379; NABTT-9809; JHOC-NABTT-9809
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2003-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma

INTERVENTIONS:
Drug: incyclinide

SUMMARY:
RATIONALE: COL-3 may stop the growth of brain tumors by stopping blood flow to the tumor.

PURPOSE: Phase I/II trial to study the effectiveness of COL-3 in treating patients who have progressive or recurrent brain tumors following radiation therapy or chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, dose limiting toxicity, and safety profile of oral COL-3 alone or when combined with anticonvulsants known to be metabolized by CYP450 in patients with progressive or recurrent high grade anaplastic astrocytoma, anaplastic oligodendroglioma, or glioblastoma multiforme.
* Define the pharmacokinetics and pharmacodynamics of COL-3 on this schedule and determine the effects of hepatic enzyme inducing drugs, such as anticonvulsants, on the pharmacokinetics.
* Determine the response rate, disease free survival, and survival in patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study of COL-3. Patients are stratified by anticonvulsant (anticonvulsants that cause induction of CYP450 vs anticonvulsants that cause modest or no induction of CYP450 or no anticonvulsant).

* Phase I: Patients receive oral COL-3 daily. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of COL-3 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

* Phase II: Patients receive oral COL-3 daily at the MTD from the phase I portion of this study.

Patients are followed every 2 months until death.

PROJECTED ACCRUAL: A total of 15-18 patients will be accrued for phase I of the study and a total of 35 patients will be accrued for phase II of the study at a rate of 3 patients per month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven high grade glioma that is progressive or recurrent following radiotherapy or chemotherapy

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Prior low grade glioma that has progressed to high grade glioma following radiotherapy and/or chemotherapy allowed
* Measurable disease by MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT or SGPT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No myocardial infarction, stroke, or congestive heart failure within the past 3 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study
* No serious active infection or medical illness that would preclude compliance
* HIV negative
* No history of gastrointestinal disorders that would interfere with absorption of study drug
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or breast, or basal cell or squamous cell skin cancer
* No hypersensitivity to tetracyclines or its derivatives

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent filgrastim (G-CSF)

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks since prior nitrosoureas) and recovered
* No more than 2 prior chemotherapy regimens

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior large field radiotherapy (greater than 20% of total bone marrow)
* At least 3 months since other prior radiotherapy and recovered

Surgery:

* No prior major upper gastrointestinal surgery
* At least 14 days since other prior major surgery

Other:

* No other concurrent investigational agents
* No prolonged sun exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Z. New, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Rudek MA, New P, Mikkelsen T, Phuphanich S, Alavi JB, Nabors LB, Piantadosi S, Fisher JD, Grossman SA. Phase I and pharmacokinetic study of COL-3 in patients with recurrent high-grade gliomas. J Neurooncol. 2011 Nov;105(2):375-81. doi: 10.1007/s11060-011-0602-9. Epub 2011 May 6. PMID 21547395